CLINICAL TRIAL: NCT07173894
Title: Randomized Control Study: The Effectiveness of Field Block (Local Anesthesia) Compared With Interscalene Block in Shoulder Surgery.
Brief Title: Effectiveness of Field Block Compared With Interscalene Block in Shoulder Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, FERAS QAWASMI, Orthopedic Surgeon, Department of Orthopedic Surgery, Hasharon Hospital, Rabin Medical Center, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HASH-ORTHO-FBvsISB-2025
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Regional Anesthesia Techniques in Shoulder Surgery
Keywords: Shoulder Surgery, Open Shoulder Surgery, Postoperative Pain, Pain Management, Regional Anesthesia, Interscalene Block
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, parallel-group comparative study designed to evaluate the effectiveness and safety of a novel Shoulder Field Block (SFB) technique performed by an orthopedic surgeon versus the standard Interscalene Brachial Plexus Block (ISB) performed by an anesthesiologist in patients undergoing shoulder surgery.
  Patients will be randomized in a 1:1 ratio to receive either the SFB or ISB technique prior to surgery. The field block is performed intraoperatively after general anesthesia using anatomical landmarks, whereas ISB is performed preoperatively using ultrasound guidance. Both groups will receive the same general anesthetic protocol and standardized multimodal perioperative analgesia.
  Pain scores, opioid use, complications, and satisfaction will be assessed over a 48-hour postoperative period. The study aims to assess whether the field block is non-inferior to ISB in terms of pain control while offering potential advantages such as fewer complications
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder Field Block by Orthopedic Surgeon (Experimental): Participants in this arm will receive a shoulder field block performed by the orthopedic surgeon using anatomical landmarks after induction of general anesthesia. The block targets the suprascapular, axillary, and lateral pectoral nerves using a tumescent local anesthetic mixture of lidocaine with epinephrine, bupivacaine, and saline to provide intraoperative and postoperative analgesia. This novel technique aims to provide effective pain relief with fewer side effects compared to the standard interscalene brachial plexus block.
  Interventions: Procedure: Shoulder Field Block by Orthopedic Surgeon
- Interscalene Block by Anesthesiologist (Active Comparator): Participants in this arm will receive a standard interscalene brachial plexus block performed by an anesthesiologist under ultrasound guidance before surgery. This block anesthetizes the upper brachial plexus nerves to provide effective intraoperative and postoperative analgesia for shoulder surgery. It is the current standard of care but may be associated with side effects such as diaphragmatic paralysis and arm weakness.
  Interventions: Procedure: Interscalene brachial plexus block and superficial cervical plexus block

INTERVENTIONS:
Procedure: Shoulder Field Block by Orthopedic Surgeon — For Shoulder Field Block intervention:
  This intervention involves a regional anesthesia technique targeting the sensory nerves of the shoulder surgical field: the suprascapular, axillary, and lateral pectoral nerves. The block is performed intraoperatively by the orthopedic surgeon using anatomical landmarks after induction of general anesthesia. A mixture of lidocaine with epinephrine, bupivacaine, and saline is injected into the shoulder area to provide local anesthesia and prolonged postoperative analgesia. This technique aims to spare the phrenic nerve, potentially reducing respiratory complications associated with traditional blocks.
  Arms: Shoulder Field Block by Orthopedic Surgeon
Procedure: Interscalene brachial plexus block and superficial cervical plexus block — This intervention involves a standard interscalene brachial plexus block performed preoperatively by an anesthesiologist under ultrasound guidance. It anesthetizes the upper roots (C5-C7) of the brachial plexus to provide effective analgesia for shoulder surgery. While effective, it carries risks such as hemi-diaphragmatic paralysis, Horner's syndrome, and motor weakness of the ipsilateral arm due to spread to adjacent nerves.
  Arms: Interscalene Block by Anesthesiologist

SUMMARY:
This study will compare two different types of anesthesia used for shoulder surgery. The first method, called an interscalene block, is commonly performed by anesthesiologists and is effective for pain control but may cause side effects such as breathing problems, arm weakness, or discomfort. The second method, called a shoulder field block, is a newer technique performed by orthopedic surgeons that numbs the nerves around the shoulder without affecting breathing.

Patients scheduled for shoulder surgery will be randomly assigned to receive either the interscalene block or the shoulder field block. The main goal of the study is to find out whether the shoulder field block provides pain relief that is as effective as the interscalene block, but with fewer side effects.

Pain levels, patient satisfaction, length of hospital stay, need for pain medication, and any complications will be recorded and compared between the two groups. The results may help identify a safe and effective alternative anesthesia option for patients undergoing shoulder surgery.

DETAILED DESCRIPTION:
Regional anesthesia is widely used for shoulder surgery, most commonly with an interscalene brachial plexus block (ISB). While ISB provides effective pain relief, it is associated with side effects such as hemidiaphragmatic paralysis, breathing difficulties, Horner's syndrome, nerve injury, and rebound pain. These risks limit its use in patients with respiratory conditions, obesity, or other contraindications.

A shoulder field block (FB) is a newer approach that targets the suprascapular, axillary, and lateral pectoral nerves, which supply most of the sensation to the shoulder joint. Unlike ISB, the field block does not affect the phrenic nerve, making it a potentially safer option. Cadaveric and early clinical studies suggest that field blocks may provide effective pain relief with fewer complications, but direct comparisons with ISB in surgical patients are limited.

This randomized controlled trial will enroll 64 adult patients undergoing arthroscopic or open shoulder surgery. Patients will be randomized into two groups:

Field Block Group: Local anesthesia field block performed by an orthopedic surgeon using anatomical landmarks.

Interscalene Block Group: Standard interscalene block performed by an anesthesiologist.

The primary outcome will be postoperative pain intensity measured by a numerical rating scale (0-10) at multiple time points during the first 48 hours. Secondary outcomes include patient satisfaction, hospital length of stay, opioid consumption, complications, and unplanned medical visits due to pain.

The study hypothesis is that a shoulder field block will provide pain relief that is non-inferior to an interscalene block, while reducing side effects and improving patient satisfaction. If effective, this technique could offer a practical alternative that can be safely performed by orthopedic surgeons, expanding anesthesia options for shoulder surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Scheduled for arthroscopic or open shoulder surgery

Exclusion Criteria:

* Prior surgery or trauma to the shoulder
* Revision shoulder surgery
* Fibromyalgia
* Pregnancy
* Contraindications to regional anesthesia (e.g., allergy to local anesthetics, coagulopathy, local site infection)
* Preexisting neuropathy or myopathy of the surgical limb
* History of chronic opioid use
* Cognitive impairment or inability to understand pain scoring systems (e.g., dementia)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity measured by Numerical Rating Scale (NRS) | From 1 hour postoperative until 48 hours after surgery
  Pain intensity will be assessed using an 11-point Numerical Rating Scale (NRS) where 0 = no pain and 10 = worst pain imaginable. Measurements will be taken at 1 hour postoperatively in the Post-Anesthesia Care Unit (PACU), at discharge from PACU, and at 6, 12, 24, and 48 hours after surgery. This outcome evaluates the effectiveness of the Shoulder Field Block compared to the Interscalene Block in controlling postoperative pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin medical center- Hasharon hospital, Petah Tikva, Central District, Israel

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the article, including data tables, will be shared. This includes pain scores (NRS), opioid consumption, complication rates, and patient satisfaction scores.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documentation will be available beginning 6 months after publication and will remain available for up to 3 years following the publication date.
Access Criteria: Qualified researchers with a methodologically sound proposal may request access to the data. Requests should be submitted to the principal investigator via institutional email. Data will be provided through a secure data-sharing platform, after approval of a data use agreement.
URL: https://clinicaltrials.gov

REFERENCES:
- [Background] Auyong DB, Hanson NA, Joseph RS, Schmidt BE, Slee AE, Yuan SC. Comparison of Anterior Suprascapular, Supraclavicular, and Interscalene Nerve Block Approaches for Major Outpatient Arthroscopic Shoulder Surgery: A Randomized, Double-blind, Noninferiority Trial. Anesthesiology. 2018 Jul;129(1):47-57. doi: 10.1097/ALN.0000000000002208. PMID 29634491